CLINICAL TRIAL: NCT02515695
Title: Bioavailability, Pharmacokinetic and Pharmacodynamic Profile of Interferon Beta-1a (Bioferon®) Administered i.v. and s.c. as Single Doses to Healthy Subjects
Brief Title: Phase I BP Interferon (IFN) Beta-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: BioPartners GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Jérôme Biollaz, MD, Chief Physician, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE 92/05; 2005DR1151 (Registry Identifier: Swissmedic)
Record Dates: First submitted 2015-07-24; First posted 2015-08-05 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.5 MIU i.v. and 1.5 MIU s.c. (Experimental): All 12 subjects participated in 4 periods, receiving 4 different doses of interferon beta-1a from 2 of the 4 possible pairs of treatments.
  The number of treatment sequences was limited to 6 and the subjects were randomized among the 6 sequences, as one male and one female per sequence. Thus 6 subjects received each dose. The washout period between two injections (Day 1 of subsequent periods) was of 7 days or more.
  Interventions: Drug: Interferon beta-1a
- 1 MIU i.v. and 3 MIU s.c. (Experimental): All 12 subjects participated in 4 periods, receiving 4 different doses of interferon beta-1a from 2 of the 4 possible pairs of treatments.
  The number of treatment sequences was limited to 6 and the subjects were randomized among the 6 sequences, as one male and one female per sequence. Thus 6 subjects received each dose. The washout period between two injections (Day 1 of subsequent periods) was of 7 days or more.
  Interventions: Drug: Interferon beta-1a
- 2 MIU i.v. and 6 MIU s.c. (Experimental): All 12 subjects participated in 4 periods, receiving 4 different doses of interferon beta-1a from 2 of the 4 possible pairs of treatments.
  The number of treatment sequences was limited to 6 and the subjects were randomized among the 6 sequences, as one male and one female per sequence. Thus 6 subjects received each dose. The washout period between two injections (Day 1 of subsequent periods) was of 7 days or more.
  Interventions: Drug: Interferon beta-1a
- 4 MIU i.v. and 12 MIU s.c. (Experimental): All 12 subjects participated in 4 periods, receiving 4 different doses of interferon beta-1a from 2 of the 4 possible pairs of treatments.
  The number of treatment sequences was limited to 6 and the subjects were randomized among the 6 sequences, as one male and one female per sequence. Thus 6 subjects received each dose. The washout period between two injections (Day 1 of subsequent periods) was of 7 days or more.
  Interventions: Drug: Interferon beta-1a

INTERVENTIONS:
Drug: Interferon beta-1a — 6 MIU/0.53 mL in pre-filled glass syringe solubilized in aqueous isotonic buffered solution
  Other Names: Bioferon®

SUMMARY:
Phase I study aiming at:

* assessing the absolute bioavailability, pharmacokinetic profile, and dose proportionality of interferon beta-1a (HSA-free solution in pre-filled syringes) after i.v. and s.c. administration as well as the pharmacodynamic profile to create the link with available surrogate markers investigated with both formulations used clinically, lyophilisate with HSA (HSA+) and solution without HSA (HSA-);
* gathering further information on safety and tolerability of interferon beta-1a over dose range,including local and systemic tolerance, body temperature, vital signs, and a battery of exploratory sickness behavior tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged between 18 and 45 years
* Weight range between 55 and 95 kg for males, 45 and 80 kg for females, providing body mass index (BMI) was between 18 and 29 kg/m2
* Absence of significant findings in the medical history and physical examination
* Absence of significant laboratory abnormalities as judged by the investigator.
* 12-lead ECG without significant abnormalities
* Negative urine drug screen

Exclusion Criteria:

* History of major renal, hepatic, immunological, haematological, gastrointestinal, genitourinary, neurological, or rheumatological disorders
* Active diseases of any type, even if mild, including inflammatory disorders and infections.
* Pregnant or lactating women or women contemplating becoming pregnant during study. Female subjects of child-bearing potential who did not practice efficient contraception during the study. A pregnancy test in blood was performed at screening and before each period with β-human chorionic gonadotropin for females of child-bearing potential. If pregnancy test was positive, the subject had to be immediately excluded from study and followed until delivery
* History of severe allergy or of asthma at any time.
* History of cardiovascular dysfunction
* Hypertension
* Sick sinus syndrome or known long QT syndrome
* Presence of QTc ￼ > 440 msec or pronounced sinus bradycardia (<40 bpm/min), even if elicited by sport
* Dark skin preventing local tolerance assessment or abnormal cutaneous reaction e.g. urticaria or papular dermographism
* Intense sport activities.
* Any clinically significant laboratory value on screening that were not within normal range on single repeat
* Positive hepatitis B & C antigen screen
* Positive HIV antibody screen or screen not performed
* Any recent acute illness or sequelae thereof which could expose the subject to a higher risk or might confound the results of the study
* Treatment in the previous three months with any drug known to have well-defined potential for toxicity to a major organ
* History of hypersensitivity to any drug if considered as serious
* History of alcohol or drug abuse
* Positive qualitative urine drug test at screening
* Use of any medication in 2 weeks prior to study and throughout study, including aspirin or other over-the-counter preparation.
* Blood (500 mL) donation or hemorrhage during the previous three months
* Participation in a clinical trial in the previous 3 months
* Smoking
* Consumption of a large quantity of coffee, tea or equivalent
* Present consumption of a large quantity of alcohol or wine or equivalent
* Psychological status which could have had an impact on subject's ability to give informed consent or behavioral tests
* Any feature of subject's medical history or present condition which, in the investigator's opinion, could confound the results of the study, complicate its interpretation, or represent a potential risk for the subject

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Composite of interferon beta-1a PK parameters | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72 [hours post-dose]
  Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-inf]) and maximum observed concentration (Cmax) following single dose administration will be assessed. Mean residence time (MRT), half-life of elimination (t1/2), clearance (CL), and volume of distribution at steady-state (Vss) will be calculated.
Composite of interferon beta-1a PD markers | 0, 6, 12, 24, 48, 72, 96, 120, 168 [hours post-dose]
  Serum concentration of three surrogate markers (neopterin and beta2-microglobulin and 2',5' OAS) will be measured

SECONDARY OUTCOMES:
Number of participants with adverse events (AE)/serious adverse event (SAE) as a measure of safety and tolerability | Up to Day 7
  AE/SAE will be collected from the start of study treatment and until the follow-up visit
Composite of local reactions as a measure of local tolerance | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 24 [hours post-dose] and then daily if needed until Day 5 or longer until resolution in case of local reaction
  Any local symptoms rated as moderate (grade 3 for i.v. and 2 for s.c.) or severe (grade 4 and 5 for i.v.; grade 3 for s.c.) will be reported as an adverse event. The subjective painful sensation following injection of the drug will be assessed using a visual analogue scale (VAS).
Composite of clinical laboratory tests as a measure of safety and tolerability | Screening and 0, 24 [hours post-dose]
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis
Composite of vital signs as a measure of safety and tolerability | Screening and 0, 1, 2, 4, 6, 8, 10, 12, 24 [hours post-dose]
  Vital signs will include body temperature, blood pressure and heart rate
Sickness behavior assessment | 0, 2, 4, 6, 8, 10, 12 [hours post-dose]
  Nine parameters will be recorded (Spontaneous movement, Ambient temperature preference, Subjective feelings, Investigator's feelings, Intellectual concentration ability, Hunger/anorexia,Thirst, Paracetamol consumption, Menthol tablet consumption)
Electrocardiogram (ECG) as a measure of safety and tolerability | Screening and 0, 8 [hours post-dose]
  Twelve-lead ECG will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Biollaz, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois

REFERENCES:
- [Derived] Perrottet N, Brunner-Ferber F, Grouzmann E, Spertini F, Biollaz J, Buclin T, Widmer N. Biases affecting injected doses of an experimental drug during clinical trials. Trials. 2016 Jul 16;17(1):321. doi: 10.1186/s13063-016-1463-5. PMID 27423899